CLINICAL TRIAL: NCT04252248
Title: Decitabine Treatment in HPV-Induced Anogenital and Head and Neck Cancer Patients After Radiotherapy or as Novel Late Salvage (DERANO)
Brief Title: Decitabine Treatment in HPV-Induced Anogenital and Head and Neck Cancer Patients After Radiotherapy or as Novel Late Salvage
Acronym: DERANO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Organizational reasons
Sponsor: University Hospital Heidelberg (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other); Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Principal Investigator, Juergen Debus, Medical Director for the Department of Radiation Oncology and Radiation Therapy, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2014-0250
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer; Anogenital Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum 1 (Experimental): Patients having received standard, definitive chemoradiotherapy according to current, national guidelines with curative intent and being at high risk for disease recurrence (patients are considered at high risk if they display a positive nodal status of their cancer (anogenital HPV-induced tumor) or if the tumor is locally advanced and/or if they display a positive nodal status with extracapsular extension (head and neck HPV-induced tumor). Study therapy (as additional therapy to standard chemoradiation) will start after a time interval of 6-8 weeks after finishing chemoradiotherapy
  Interventions: Drug: Dacogen
- Stratum 2 (Experimental): Patients with non-curative and progressive disease having received all standard, national approved systemic therapies (according to current, national guidelines with regard to the specific tumor entity), and/or presently not eligible for a respective therapy, and/or refused respective therapy. Study treatment thereby represents a potential palliative, "last-line" systemic therapy option (late salvage).
  Interventions: Drug: Dacogen

INTERVENTIONS:
Drug: Dacogen — Intravenous (i.v.) infusion of 20 mg/m2 over 1 hour repeated daily for 5 days starting on day 1. Single repetition of cycle on day 29.

SUMMARY:
Open-label, single-center phase I study to evaluate first signs of efficacy and to confirm the safety and tolerability of a decitabine safe-dose treatment in two strata of patients with HPV induced anogenital and head and neck cancers (Stratum 1: patients with high rist for disease recurrence; Stratum 2: patients with failure of standard therapy). The study is expected to enroll 18 patients overall (9 patients in each stratum).

The duration of the trial for each patient is expected to be 6 months (two 28 day cycles of study treatment plus four months of additional follow-up). The overall duration of the trial is expected to be approximately 42 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting all of the following criteria will be considered for admission to the trial: Patients with an HPV-induced (will be assumed if both HPV DNA and immunohistochemical overexpression of p16INK4a is detected in tumor tissue) cancer of the

* anus
* vulva
* vagina
* uterine
* cervix
* penis or
* oropharynx/oral cavity and

  * Stratum 1: Patients having received standard, definitive chemoradiotherapy according to current national guidelines with curative intent and being at high risk for disease recurrence (patients are considered at high risk if they display a positive nodal status of their cancer (anogenital HPV-induced tumor) or if the tumor is locally advanced and/or if they display a positive nodal status with extracapsular extension (head and neck HPV-induced tumor). Study therapy (as additional therapy to standard chemoradiation) will start after a time interval of 6-8 weeks after finishing chemoradiotherapy.
  * Stratum 2: Patients with non-curative and progressive disease having received all standard, national approved systemic therapies (according to current, national guidelines with regard to the specific tumor entity), and/or presently not eligible for a respective therapy, and/or refused respective therapy. Study treatment thereby represents a potential palliative, "last-line" systemic therapy option (late salvage).
* Ability of patient to understand character and individual consequences of the clinical trial
* Postmenopausal or evidence of non-childbearing status. For women of childbearing potential: negative urine pregnancy test at baseline and highly effective forms of contraception (see 6.5) in place thereafter as well as confirmed negative urine pregnancy test prior to treatment on day 1 of every cycle and at end of treatment period Evidence of childbearing potential is defined as:

  * Fertile, following menarche and until becoming post-menopausal unless permanently sterile Postmenopausal or evidence of non-childbearing status is defined as: o Amenorrheic for 1 year or more without an alternative medical cause following cessation of exogenous hormonal treatments PLUS Follicle stimulating hormone (FSH) levels in the postmenopausal range in women not using hormonal contraception or hormonal replacement therapy
  * Surgical sterilisation (bilateral oophorectomy, hysterectomy or bilateral salpingectomy) A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.
* Female patients of child bearing potential and male patients with partners of child bearing potential, who are sexually active, must agree to the use of highly effective forms of contraception. This should be started from the signing of the informed consent and continue throughout period of taking study treatment and for 6 months (female study participants)/ 3 months (male study participants) after last dose of study drug.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study (must be given before enrolment in the trial)
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Patients presenting with any of the following criteria will not be included in the trial:

* Age <18 years
* Grade 3 neutropenia with Neutrophiles < 1/nl, thrombocytopenia with thrombocytes < 50/nl and/ or anemia with Hgb <8.0 g/dL
* Active infections requiring anti-infective treatment
* Bleeding disorders (e.g. Hemophilia, von Willebrandt disease, congestive deficiency of any coagulation factor (e.g. factor V, X), Immune thrombocytopenia (ITP) thrombocytopathies (e.g. Bernard-Soulier-syndrome drug induced bleeding disorders
* Insulin-dependent and unregulated diabetes
* Grade 3/4 renal failure with a GFR < 60 ml/min
* Liver cirrhosis Child C • History of cardiac diseases
* Pregnancy and/ or lactation • History of treatment with DNA Methyltransferase Inhibitors (DNMTs)
* Participation in other clinical trials involving another investigational agent within 4 weeks prior to first treatment of this study
* ECOG performance status >2
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* History of other malignancies (except basal cell carcinoma) in the past 5 years No patient will be allowed to enroll in this trial more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) | 56 days
  The primary objective of the study is to evaluate the safety and tolerability of decitabine treatment in two strata of patients with HPV-induced anogenital and head and neck cancer. Primary endpoint is the incidence of dose limiting toxicities (DLT) during the first two cycles of study treatment (up to day 56). DLT will be assessed and managed independently for both strata.

SECONDARY OUTCOMES:
Overall Response Rate | 6 months
  The Overall Response Rate (or Objective Response Rate) is defined as the proportion of patients achieving a complete (CR) or partial (PR) response in their overall response assessment according to RECIST v1.1 measured at the 6 months staging vs baseline.
Disease Control Rate (DCR) | 6 months
  The Disease Control Rate (DCR) is defined as the proportion of patients achieving stable disease or a better outcome (CR, PR, SD) in their overall response assessment according to RECIST v1.1 measured at the 6 months staging vs baseline.
Quality of Life | week 3, 5, 8 and 24
  Quality-of-Life (QoL) will be assessed by the EORTC Quality of Life Core Questionnaire (QLQ30), supplemented by information on self-assessed concomitant diseases and demographics. QoL will be assessed at baseline, and at week 3, 5, 8 and 24 (EOS)
Overall Survival (OS) | from admission until Last Patient Last Visit (LPLV), assessed ≥ 6 months
  OS is defined as the time from admission to the study until death from any cause. Patients who are alive at the end of the study are censored on the day of last contact.
Progression-free Survival (PFS) | from admission until Last Patient Last Visit (LPLV), assessed ≥ 6 months
  PFS is defined as the time from admission to the study until progression of disease or death from any cause, whichever occurs first. Patients who are alive and did not have progression of disease at the end of the study are censored on the day of last contact.
Overall Response Rate | 3 months
  The ORR-3m is defined as the proportion of patients achieving a complete (CR) or partial (PR) response in their overall response assessment according to RECIST v1.1 measured at the 3 months staging vs baseline.
Disease Control Rate | 3 months
  The DCR-3m is defined as the proportion of patients achieving stable disease or a better outcome (CR, PR, SD) in their overall response assessment according to RECIST v1.1 measured at the 3 months staging vs baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof. Dr. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- UKHD, Klinik für RadioOnkologie und Strahlentherapie, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes